CLINICAL TRIAL: NCT01512602
Title: Efficacy of Dialectical Behavior Therapy in Patient With Self Harming Behavior and Traits Within the Spectrum of Borderline Personality Disorder.
Brief Title: Efficacy of Dialectical Behavior Therapy Versus CAMS-informed Supportive Psychotherapy on Self Harming Behavior
Acronym: DiaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Lundbeck Foundation (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Merete Nordentoft, Professor, MD, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RHP-DiaS-002
Record Dates: First submitted 2011-12-21; First posted 2012-01-19 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Borderline Personality Disorder; Suicide
Keywords: Borderline Personality Disorder traits; Suicide prevention; Self-harm; Dialectical Behavior Therapy; DBT; Collaborative Assessment and Management of Suicidology; CAMS
MeSH Terms: conditions — Borderline Personality Disorder; Suicide; Suicide Prevention; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dialectical Behavior Therapy DBT (Active Comparator): 16 weeks DBT-treatment
  Interventions: Behavioral: DBT
- CAMS (Active Comparator): Collaborative Assessment and Management of Suicidality, CAMS-informed supportive psychotherapy
  Interventions: Behavioral: CAMS

INTERVENTIONS:
Behavioral: DBT — 16 weeks DBT treatment
  Arms: Dialectical Behavior Therapy DBT
Behavioral: CAMS — CAMS-informed psychotherapy
  Arms: CAMS

SUMMARY:
Purpose: The purpose of this study is to investigate the efficacy of Dialectical Behavior Therapy (DBT) versus CAMS (Collaborative Assessment and Management of Suicidality) -informed supportive psychotherapy on the risk of self-harm acts and suicide attempts in patients with self behavior and personality traits within the spectrum of borderline personality disorder.

Hypothesis: The hypothesis is 16 weeks of treatment with Dialectical Behavior Therapy (DBT) after a defined manual has a higher efficacy than CAMS-informed supportive psychotherapy on self-harm acts, suicide attempts, suicidal ideation, depressive symptoms, impulsiveness and consumption of hospital services in patients with symptoms within the spectrum of borderline personality disorder (BDP).

Method: The investigators will include 160 patients in the randomized trial to investigate whether 16 weeks of DBT-treatment as a higher efficacy than CAMS-informed supportive psychotherapy on the risk of self-harm acts and suicide attempts in patients with self-harm behavior and personality traits within the spectrum of borderline personality disorder. The trial will meet strict criteria for high quality randomized trials, and will hopefully help to establish evidence for the treatment of this patient group at higher risk of later suicide. There will be performed follow up interviews after 16 weeks, 28 weeks and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* Newly suicide attempt within one month of the inclusion date.
* A minimum of two characteristics in the DSM-IV Borderline Personality Disorder (BPD)
* Informed consent.

Exclusion Criteria:

* Severe depression.
* Bipolar disorder.
* Psychosis within the schizophrenic spectrum.
* Anorexia Nervosa.
* Substance abuse.
* Mental retardation.
* Dementia.
* Lack of informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of repeated self-harming acts including suicide attempts (change in number of self-harming acts). | Week 0 (baseline), 17, 28, 52.
  This information will be obtained as self-reported and through journal entries.How many acts how has taken place between the different time points in the trial (week 0, 17,28, and 52) to actually quantify the self-harming acts in order to find out if the treatment in the two arms can decrease the numbers of self-harming acts, also long term effect (week 52).

SECONDARY OUTCOMES:
Depressive symptoms | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by HDRS-17 and BDI.
Impulsivity | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by Barratts Impulsivity Scale (BIS-11)
Consumptions of services in hospital care. | After treatment period (16 weeks), Week 28 and 52 after inclusion
  Register based information: Contact with hospital contact with code 4 (self-harm act), or suicide attemp X60-X84, or poisioning by weak analgesia (T39), hypnotics (T52), or psychothopic drugs (T43). Vital status, causes of death, use of bed days and outpatients services.
Suicidal ideation | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by Beck's Suididal Ideation Scale (SSI-21)
Severity of borderline personality disorder symptoms. | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by Zanarini Borderline Personality Scale.
Anger | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by State Trait Anger Scale.
Hopelessness | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion.
  Measured by Becks Hopelessness Scale.
Self Esteem | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion
  Measured by Rosenbergs Self esteem Scale (RSE).
Suicide related behavior. | Assessed at baseline, after treatment period (16 weeks), Week 28 and 52 after inclusion.
  Measured by Suicide Attempt Self Injury Interview (SASII) and Beck's suicide intent Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Services, Research Unit, Bispebjerg, Copenhagen NV., Denmark

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793
- [Derived] Andreasson K, Krogh J, Wenneberg C, Jessen HK, Krakauer K, Gluud C, Thomsen RR, Randers L, Nordentoft M. EFFECTIVENESS OF DIALECTICAL BEHAVIOR THERAPY VERSUS COLLABORATIVE ASSESSMENT AND MANAGEMENT OF SUICIDALITY TREATMENT FOR REDUCTION OF SELF-HARM IN ADULTS WITH BORDERLINE PERSONALITY TRAITS AND DISORDER-A RANDOMIZED OBSERVER-BLINDED CLINICAL TRIAL. Depress Anxiety. 2016 Jun;33(6):520-30. doi: 10.1002/da.22472. Epub 2016 Feb 8. PMID 26854478
- [Derived] Andreasson K, Krogh J, Rosenbaum B, Gluud C, Jobes DA, Nordentoft M. The DiaS trial: dialectical behavior therapy versus collaborative assessment and management of suicidality on self-harm in patients with a recent suicide attempt and borderline personality disorder traits - study protocol for a randomized controlled trial. Trials. 2014 May 29;15:194. doi: 10.1186/1745-6215-15-194. PMID 24885904